CLINICAL TRIAL: NCT07332663
Title: Exploratory Study on the Treatment of Relapsed and Refractory B-cell Malignant Tumors With WGb-0301 Injection
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19 CAR-T for B cell cancer
Record Dates: First submitted 2025-12-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: B Cell Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WGb-0301 injection (Experimental)
  Interventions: Drug: WGb-0301 injection

INTERVENTIONS:
Drug: WGb-0301 injection — WGb-0301 injection

SUMMARY:
Malignant hematological tumors mainly derived from adult B cells are mainly acute lymphoblastic leukemia (ALL) and non Hodgkin lymphoma (NHL). Overall, although existing therapies have significantly improved the survival rates of most patients, the treatment of relapsed/refractory patients still faces significant challenges. CD19 is one of the most clinically valuable targets for B-cell malignant hematological tumors.

The advent of COVID-19 vaccine has brought LNP mRNA technology into the public's view. After years of development, it not only shines brilliantly in COVID-19 vaccine, but also is widely used in the treatment and exploration of cancer, rare diseases and other fields. The core of LNP mRNA technology targeting CD19 is to encapsulate the mRNA encoding specific proteins in lipid nanoparticles and deliver them to the body through intravenous or intramuscular injection.

The experimental drug WGb-0301 injection is a CD19 based messenger RNA (mRNA) therapeutic mRNA drug, formed by loading mRNA onto lipid nanoparticles (LNP). WGb-0301 injection has demonstrated efficient B-cell clearance activity and good safety in non clinical settings, supporting further clinical exploration in B-cell malignancies. It is expected to provide an innovative, safe, and accessible immunotherapy for B-cell malignancies, bringing better clinical benefits to more patients with B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range of 18-70 years old, gender not limited;
* 2. Expected survival time exceeds 12 weeks;
* 3. B-cell lymphoma or lymphocytic leukemia diagnosed with CD19+, with no standard treatment options recommended according to guidelines and meeting the corresponding frontline treatment line requirements;
* 4. There are assessable lesions (applicable only to lymphoma patients);
* 5. The physical fitness status score of the Eastern Cancer Collaboration Group (ECOG) is 0 or 1 point;
* 6. The main organ functions well and the relevant examination indicators meet the corresponding requirements;
* 7. Male and female patients of appropriate age must use reliable methods of contraception before entering the trial, during the research process until 30 days after discontinuation of medication; Reliable contraceptive methods will be determined by the primary researchers or designated personnel;
* 8. Those who can understand this experiment and have signed the informed consent form.

Exclusion Criteria:

* 1. Accompanied by other uncontrolled malignant tumors;
* 2. Previously received chimeric antigen receptor therapy or other transgenic T cell therapy;
* 3. Known history of HIV or hepatitis B (HBsAg positive and HBV DNA reaching the detection limit) or hepatitis C virus (anti HCV positive) infection;
* 4. Participants with a history of CNS lymphoma, malignant cells in cerebrospinal fluid, or brain metastases;
* 5. Participants with atrial or ventricular involvement;
* 6. Emergency treatment is required due to the impact of tumor masses, such as intestinal obstruction or vascular compression;
* 7. Suffering from serious diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage, poorly controlled hypertension, or other uncontrolled active diseases that hinder participation in the trial;
* 8. Unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolism events occurred within 30 days prior to enrollment. If receiving anticoagulant therapy, the treatment dose of participants must reach a stable level before enrollment;
* 9. For those who have been using immunosuppressants for a long time after organ transplantation, except for recent or current inhaled corticosteroid therapy;
* 10. Any pregnant or breastfeeding woman, or participant who plans to conceive during or within 18 months after treatment;
* 11. Within 14 days prior to enrollment, there is an active or uncontrollable infection that requires systemic treatment (excluding simple urinary tract infections or upper respiratory tract infections);
* 12. The researcher believes that there are any other factors that are not suitable for the study participants to enter this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) and its incidence rate | Within 90 days after the initial treatment
Maximum tolerated dose (MTD) or optimal biological dose (OBD) | Through study completion, an average of 2 year

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 2 year
Disease control rate (DCR) | Through study completion, an average of 2 year
Duration of response (DoR) | From the date of the first PR/CR to the date of the first confirmation of progress or death for any reason
Progression free survival (PFS) | From the date of initial treatment until the first confirmation of progression or death for any reason